CLINICAL TRIAL: NCT02495129
Title: A Three-part, Partially Open Label and Double-blind, Randomized Study to Assess the Pharmacodynamic Effects, Safety, Tolerability and Preliminary Efficacy of VAY736 in Patients With Primary Sjögren's Syndrome Using [Zr-89]-Rituximab PET/CT
Brief Title: Study of Pharmacodynamic Effects of VAY736 in Patients With Primary Sjögren's Syndrome
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAY736X2103
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-02

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Primary Sjögren's syndrome; Sicca syndrome; Salivary glands; Positron Emission Tomography; B cell depletion
MeSH Terms: conditions — Sjogren's Syndrome | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- VAY736 lower dose (Experimental): 12 evaluable patients will be enrolled and randomized (at a ratio of 1:1) to receive either a lower dose or a higher dose of the study drug (VAY736)
  Interventions: Drug: VAY736 lower dose
- VA736 higher dose (Experimental): 12 evaluable patients will be enrolled and randomized (at a ratio of 1:1) to receive either a lower dose or a higher dose of the study drug (VAY736)
  Interventions: Drug: VAY736 higher dose

INTERVENTIONS:
Drug: VAY736 lower dose — Patients will receive a total number of 3 monthly subcutaneous injections with the lower dose of VAY736
  Arms: VAY736 lower dose
Drug: VAY736 higher dose — Patients will receive a total number of 3 monthly subcutaneous injections with the higher dose of VAY736
  Arms: VA736 higher dose

SUMMARY:
This study consists of three consecutive parts. Part 1 in primary Sjögren's syndrome (pSS) patients (n=2-6) and Part 2 in healthy voluteers (n=3) are feasibility studies to assess if the selected [Zr-89]-rituximab PET/CT method is a valid method to assess B cells in salivary glands of pSS patients. In Part 1 and Part 2 no IMP will be applied to the subjects. In Part 3, pSS patients (n=12) will receive the IMP, VAY736. Posted information will be focused on Part 3.

The overarching purpose of this study is to test a new drug (VAY736) for the treatment of pSS. In pSS, the salivary glands (the glands that produce saliva) and other organs are affected by inflammation. A certain type of white blood cells called B cells prominently infiltrate the salivary glands in pSS, whereas they are not present in healthy salivary glands. Scientific evidence suggests that B cells may be involved in the disease process in pSS and that eliminating B cells may benefit patients with pSS. This study will test a new imaging method and a new treatment for pSS. Both the imaging method and the treatment are specific for B cells.

ELIGIBILITY:
Part 1 and 3:

Inclusion Criteria:

* Fullfilled consensus criteria for primary Sjögren's syndrome
* Patients must have elevated serum levels for some Sögren Syndorme specific parameters such as antinuclear antibodies (ANA), rheumatoid factor (RF) etc.

Exclusion Criteria:

* Patients that are suffering from Secondary Sjögren's syndrome.
* Patients previously treated with monoclonal antibody treatments such as rituximab, infliximab, adalimumab, etc.

Part 2

Inclusion criteria:

- healthy male and female people 18-75 years of age

Exclusion criteria:

* Use of other investigational drugs at the time of enrollment
* Exposure to a sizeable degree of radiation (≥ 5 mSv) in an investigational research study in the past year prior to this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Part 1: To determine the feasibility of measuring major salivary gland infiltrating B cells in pSS patients using [Zr- 89]rituximab PET/CT imaging | Part 1: 4 weeks
  Part 1: PET/CT imaging of pSS major salivary gland 3, 6 and 9 days after i.v. injection with [Zr- 89]rituximab
Part 2: To define the normal range of PET/CT imaging values for major salivary gland tissue, cervical lymph nodes and spleen in healthy volunteers with [Zr-89]-rituximab | Part 2: 4 weeks
  Part 2: PET/CT imaging of healthy volunteers' major salivary gland, cervical lymph nodes and spleen on optimal time point after i.v. injection with [Zr-89]-rituximab (e.g. 3 days after injection)
Part 3: To compare the effect of two different VAY736 s.c. dose regimes on salivary gland-infiltrating B cells in pSS patients, using [Zr-89]-rituximab PET/CT imaging | Part 3: 12 weeks
  Part 3: PET/CT imaging of pSS tissues on optimal time point after i.v. injection with [Zr-89]-rituximab, at baseline and 12 weeks after the start of VAY736 treatment

SECONDARY OUTCOMES:
Safety of multiple s.c. dosing of VAY736 in pSS patients as measured by safety assessments | 12 weeks
  AEs, vital signs, ECGs, safety laboratory parameters (Hematology, Biochmistry, Urinalysis)
To asses the pharmacokinetiks of VAY736 in pSS patients | 12 weeks
  Multiple s.c. dose VAY736 PK parameter - Area under the curve (AUC)
To assess the pharmacokinetiks of VAY736 in pSS patients | 12 weeks
  Multiple s.c. dose VAY736 PK parameter - Trough concentrations after multiple dose
Assess the pharmacodynamic effect of VAY736 on circulating CD19+ B-cells in pSS | 12 weeks
  Multiple s.c. dose VAY736 PD parameter - depletion of B cells
Asses effect of two different VAY736 dose levels on target tissue structure and function in pSS | 12 weeks
  Assess size of spleen and cervical lyph nodes by PET/CT imaging and ultrasound-aided size measurements
Asses effect of two different VAY736 dose levels on target tissue structure and function in pSS | 12 weeks
  Assess salivary glands size and echostructure by ultrasound
Asses effect of two different VAY736 dose levels on target tissue structure and function in pSS | 12 weeks
  Assess salivary gland function (quantitative) by salivary flow (stimulated and unstimulated)
Asses effect of two different VAY736 dose levels on target tissue structure and function in pSS | 12 weeks
  Assess lacrimal gland function by Schirmer's test
To evaluate the effect of two different VAY736 dose levels (s.c. q4w) on pSS disease activity | 12 weeks
  Assess the change in the EULAR Sjögren'sSyndrome Disease Activity Index (ESSDAI).
To evaluate the effect of on self-reported outcomes in pSS patients | 12 weeks
  Multidimensional Fatigue Inventory (MFI-20); the short form 36 health Survey (SF-36); EULAR Sjögren's Syndorm Patient Reported Intensity (ESSPRI)
To evaluate the change in the physician global assessment of patients's overall disease activity | 12 weeks
  Physician's visual anaglog scale (VAS)
To evaluate the change in the patients global assessment of their disease activity | 12 weeks
  Patient's visual analogue scale (VAS)
To assess the immunogenicity of VAY736 | 12 weeks
  Anti-VAY736 antibodies
To assess the immunogenicity of a micodose of rituximab | 25 weeks
  Anti-rituximab antibodies
To asses the pharmacokinetiks of VAY736 in pSS patients | 12 weeks
  Multiple s.c. dose VAY736 PK parameter - Cmax
To asses the pharmacokinetiks of VAY736 in pSS patients | 12 weeks
  Multiple s.c. dose VAY736 PK parameter - tmax
To asses the pharmacokinetiks of VAY736 in pSS patients | 12 weeks
  Multiple s.c. dose VAY736 PK parameter - half live (t1/2)